CLINICAL TRIAL: NCT02767934
Title: A Phase II Study of Anti-PD-1 Antibody (MK-3475; Pembrolizumab) for the Treatment of Minimal Residual Disease in Adults With Acute Lymphoblastic Leukemia
Brief Title: Pembrolizumab in Treating Minimal Residual Disease in Patients With Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of efficacy
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9458; NCI-2016-00602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9458 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1016006 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-06

CONDITIONS: B Acute Lymphoblastic Leukemia; Minimal Residual Disease; Recurrent Acute Lymphoblastic Leukemia; T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients achieving complete MRD response may receive up to 1 additional year of treatment at the discretion of the investigator.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating small amounts of cancer cells that remain after attempts to remove the cancer has been made in patients with acute lymphoblastic leukemia. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of pembrolizumab in minimal residual disease (MRD)-positive acute lymphoblastic leukemia (ALL).

SECONDARY OBJECTIVES:

I. To describe the toxicity profile of pembrolizumab in patients with previously-treated ALL.

II. To gain a preliminary assessment of how MRD response translates into relapse-free and overall survival.

EXPLORATORY OBJECTIVES:

I. To compare disease assessments by multiparameter flow cytometry (MFC) and polymerase chain reaction (PCR) to a newly-developed and more sensitive next generation sequencing (NGS)-based platform.

II. To correlate response to pembrolizumab to immunologic markers in peripheral blood and bone marrow specimens.

III. To evaluate if treatment with pembrolizumab has a measurable impact on hematopoietic engraftment and graft-vs-host disease (GVHD) in patients who subsequently undergo allogeneic hematopoietic cell transplantation (HCT).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients achieving complete MRD response may receive up to 1 additional year of treatment at the discretion of the investigator.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a diagnosis of ALL of either B-cell, T-cell, or mixed (i.e., B/T lineage)
* Be willing and able to provide written informed consent for the trial
* Presence of MRD (defined as < 5% blasts in the bone marrow by morphologic assessment and no clinically-apparent extramedullary disease but with quantifiably-measurable disease as assessed by either MFC or PCR) under any of the following circumstances:

  * MRD persistence >= 11 weeks after the start of initial therapy
  * MRD persistence >= 2 weeks after the start of salvage therapy, or
  * MRD reappearance at any time
* For patients with Philadelphia chromosome positive (Ph+) disease, have previously received treatment with >= 1 Abelson (ABL) kinase inhibitor (e.g., imatinib, dasatinib, etc.) or are ineligible for such treatment
* Have previously received or are ineligible for treatment with blinatumomab; ineligibility will include (but not be limited to) cluster of differentiation 19 (CD19)-negative disease, denial of insurance coverage, physician discretion, and/or patient refusal
* Be willing to provide tissue from a newly obtained bone marrow aspirate and/or biopsy; newly-obtained is defined as a specimen obtained up to 28 days prior to initiation of treatment on day 1; subjects for whom newly-obtained samples cannot be provided (e.g., inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the principal investigator (PI)
* Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,000 /mcL (performed within 10 days of treatment initiation)
* Hemoglobin >= 8 g/dL (performed within 10 days of treatment initiation)
* Platelets >= 50,000 /mcL (performed within 10 days of treatment initiation)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min/1.73 m^2 for subject with creatinine levels > 1.5 X institutional ULN (performed within 10 days of treatment initiation) (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 ULN (performed within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 3 days prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational new drug and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active bacillus tuberculosis (TB)
* Has a known hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy or with hematologic toxicity that has recovered to levels above that stated in inclusion criterion are an exception to this criterion and may qualify for the study if all other inclusion/exclusion criteria are met
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention (i.e., =< grade 1 or at baseline) prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) leukemia and/or leukemic meningitis; subjects with previously treated CNS leukemia may participate provided they are stable (e.g., without evidence of active disease by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline) and have no evidence of leukemic blasts on analysis of cerebrospinal fluid (CSF)
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has previously received an allogeneic hematopoietic cell transplant, unless the following criteria are met:

  * Detection of MRD occurred >= 21 days from stem cell infusion
  * No active GVHD
  * Receiving systemic steroid therapy of =< 10 mg of prednisone daily (or equivalent)
  * Has discontinued systemic immunosuppressant therapy >= 7 days prior to first dose of pembrolizumab
* Has previously received other forms of cellular immunotherapy (e.g., chimeric antigen receptor-modified [CAR] T cells), unless the following criteria are met:

  * Detection of MRD occurred >= 21 days from cell infusion
  * Any specific manifestations of cytokine release syndrome or neurologic toxicity attributable to the cellular therapy have completely resolved (i.e., < grade 1)
* Has an active infection requiring systemic therapy; antimicrobial prophylaxis will be permitted at the discretion of the treating investigator
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting from the time of consent through 120 days after the last dose of trial treatment
* Has received prior therapy with any immune checkpoint inhibitor
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface protein antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Cassaday, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Cassaday RD, Garcia KA, Fromm JR, Percival MM, Turtle CJ, Nghiem PT, Stevenson PA, Estey EH. Phase 2 study of pembrolizumab for measurable residual disease in adults with acute lymphoblastic leukemia. Blood Adv. 2020 Jul 28;4(14):3239-3245. doi: 10.1182/bloodadvances.2020002403. PMID 32692850

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Pembrolizumab for MRD in Adults with ALL
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Minimal Residual Disease Response
Description: Will be defined as percentage of evaluable subjects who achieve a complete response. Will be evaluated with a Simon two-stage optimum design.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab: Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients achieving complete MRD response may receive up to 1 additional year of treatment at the discretion of the investigator.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
Participants | 1

2. Secondary Outcome: Overall Survival
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
months | 12.7 [5.9 to 30.4]

3. Secondary Outcome: Relapse-Free Survival
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
months | 3.1 [1.2 to 30.4]

ADVERSE EVENTS:
Time Frame: From the time of consent through 30 days following cessation of treatment, an average of 3 months
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=12)
Bacteremia (acinetobacter ursingii, herbasprillum, achromobacter xylosoxidans) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=12)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT02767934/Prot_SAP_000.pdf